CLINICAL TRIAL: NCT05289284
Title: Aspects of Validity of the Single Leg Squat Test: A Cohort Study of Female Soccer Players.
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Rasmussen Barr, Associate Professor, Karolinska Institutet
Other Study IDs: Dnr 2021-05398-02
Record Dates: First submitted 2022-03-13; First posted 2022-03-21 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Functional Movement Disorders; Reproducibility of Results; Sports Medicine
Keywords: The Single Leg Squat; Discriminative validity; Female Soccer players; Sports Injury
MeSH Terms: conditions — Conversion Disorder; Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female soccer cohort: A female soccer cohort will be followed for 10 month regarding injuries
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Movement screening tests to identify deficits or poor movement quality is commonly used in soccer and other sports to assess injury, to evaluate rehabilitation goals and return to sport after injury.

Female soccer players have an increased risk of suffering a knee injury which can be related to a poor knee control. Knee control can be observed and assessed by the Single Leg Squat (SLS) test. The SLS test is reported to be reliable, but there still is an overall lack of clear evidence of the accuracy for tests used for assessing movement quality in sports medicine, and the discriminate and predictive validity of the SLS test in a female soccer cohort needs to be further investigated. It is also not clear what significance other physiological- psychosocial- and hormonal factors have for the outcome of the SLS and for injury.

The overall aim of this project is to investigate if the outcome of a visually assessed SLS test can discriminate between individuals with a previous injury in the lower extremity, and if the outcome, separate or together with physiological-, psychosocial- and hormonal factors can predict future injury in a cohort of female soccer players.

The authors hypothesises that the outcome of the SLS cannot discriminate between individuals with a previous injury in the lower extremity but that the outcome of the SLS, separate or together with physiological-, psychosocial- and hormonal factors can predict future injury in a cohort of female soccer players.

269 female soccer players (≥16 Yr.) from Damallsvenskan, Elitettan and division 1 in the area of Stockholm was enrolled in the study and baseline measurements were done during 2022-01-08 to 2022-02-21. The female soccer cohort will be followed during the season 2022 regarding injuries upcoming injuries.

DETAILED DESCRIPTION:
Movement screening tests to identify deficits or poor movement quality is commonly used in soccer and other sports to assess injury, to evaluate rehabilitation goals and return to sport after injury.

Female soccer players have an increased risk of suffering a knee injury which can be related to a poor knee control. Knee control can be observed and assessed by the Single Leg Squat (SLS) test which is one of the most commonly used clinical tests for assessing movement quality of the knee and other parts of the kinetic chain. The SLS test is reported to be reliable, but there still is an overall lack of clear evidence of the accuracy for tests used for assessing movement quality in sports medicine, and the discriminate and predictive validity of the SLS test in a female soccer cohort needs to be further investigated.

It is also not clear what significance physiological factors such as the range of ankle dorsi flexion, hip strength and psychosocial factors such as sleep, stress, anxiety and fear of avoidance have for the outcome of the SLS and for injury. Neither has hormonal factors such as self-assessed menstrual cycle, related factors and use of oral contraceptives been clarified regarding its significance in relation to the outcome of the SLS test and injury.

The overall aim of this project is to investigate if the outcome of a visually assessed SLS test can discriminate between individuals with a previous injury in the lower extremity, and if the outcome, separate or together with physiological-, psychosocial- and hormonal factors can predict future injury in a cohort of female soccer players.

* How is the outcome of a SLS test and its separate items associated to physical factors.
* Are the outcome of a SLS test and its separate items able to discriminate between players with and without previous injury in the lower extremity.
* Are the outcome of a SLS test, separate, or together with physical- (hip strength, ankle mobility), psychosocial- (stress, sleep, anxiety, fear of avoidance) and hormonal (self-assessed menstrual cycle, related factors and use of oral contraceptives) factors able to predict injury in the lower extremity measured every four weeks for10 months following the baseline measurements.

The authors hypothesises that the outcome of the SLS cannot discriminate between individuals with a previous injury in the lower extremity but that the outcome of the SLS, separate or together with physiological-, psychosocial- and hormonal factors can predict future injury in a cohort of female soccer players.

Twenty soccer teams from Damallsvenskan, Elitettan and division 1 in the area of Stockholm was contacted in order to recruit at least 200 female soccer players (≥16 Yr.). During autumn 2021 information about the study was sent out to the clubs by e-mail, and for those who wanted to participate, further written and verbal information was given. Before baseline assessment, which started 2022-01-08, information about the project was given verbally and in writing to the soccer players. Baseline assessment included physical assessments as well as psychosocial-, hormonal-, previous injury- and demographic questionnaires. Inclusion criteria was female soccer players contracted with a club in Damallsvenskan, Elitettan or division 1 for the season 2022 who was 16 years or older, and native in written and spoken Swedish. Exclusion was an ongoing injury in the lower extremity that made it impossible to perform the physical baseline assessments, or that the performance may present an additional risk for injury. The physical tests were performed at the local club by the doctoral student John Ressman. The time needed for baseline measurements per participant including physical tests and self-assessed questionnaires was approximately 15-20 minutes. In order to follow up on injuries during the soccer season 2022 a web-based questionnaire, the Oslo Sports Trauma Research Centre (OSTRC), was used. OSTRC is validated and designed to capture both injuries and overuse injuries in sports injury epidemiology. The web-based questionnaire will be sent via SurveyMonkey © every four weeks for 10 month following the baseline measurement.

ELIGIBILITY:
Inclusion Criteria:

* Female soccer players contracted with a club in Damallsvenskan, Elitettan or division 1 for the season 2022.
* Native in written and spoken Swedish.
* 16 years ol

Exclusion Criteria:

* Ongoing injury in the lower extremity that made it impossible to perform the physical baseline assessments, or that the performance may present an additional risk for injury

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Female soccer players contracted with a club in Damallsvenskan, Elitettan or division 1 for the season 2022.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Injury | 10 month
  Receiving an injury: time-loss or overuse
The Single Leg Squat | Cross sectional at baseline
  Fail/pass of the Single Leg squat

CONTACTS AND LOCATIONS:
Overall Officials: Eva Rasmussen Barr, Principal Investigator — Karolinska Institutet. Alfred Nobels Allé 23, 141 83 Huddinge
Locations (1):
- Karolinska Institutet, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
The datasets generated and/or analysed during the current study are not publicly available due to ethical regulation at the Karolinska Institute but are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Ressman J, von Rosen P, Grooten WJA, Rasmussen-Barr E. Factors associated with the Single Leg Squat test in female soccer players: a cross-sectional study. BMC Sports Sci Med Rehabil. 2024 Apr 2;16(1):76. doi: 10.1186/s13102-024-00853-1. PMID 38566260